CLINICAL TRIAL: NCT00794716
Title: Prospective Single-centre, Open-label Study to Assess the Pharmacokinetics of Cholyl-lysl-fluorescein (NRL972) in Patients with Clinical Evidence for NAFLD: Supporting the Disease Staging Into Fatty Liver Disease Versus NASH
Brief Title: PK of NRL972 in Patients with Nonalcoholic Steatohepatitis (NASH) and Non-Alcoholic Fatty Liver Disease (NAFLD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NRL972-01/2007 (FLD)
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — NRL972

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | US Export: No

ARMS (1):
- NRL972 (Experimental): 2 mg NRL972 IV
  Interventions: Drug: NRL972

INTERVENTIONS:
Drug: NRL972 — Single dose of 2 mg NRL972 administered intravenously. Total volume 5mL.
  Other Names: cholyl-lysyl-fluorescein

SUMMARY:
This study is to evaluate the predictive value of NRL972 pharmacokinetics in the diagnosis of steatohepatitis using fatty liver disease as the comparator group. In addition, the sensitivity and specificity of NRL972 pharmacokinetics as a diagnostic tool will be compared to results from the standard laboratory tests, elastography, tests of metabolic markers and serum fibrosis markers frequently used in the evaluation of clinically predicted NAFLD patients. Patients will be included if they have clinical evidence of fatty liver disease and have been referred to the clinic for a diagnostic work-up, including a liver biopsy, blood tests and scans of the liver.

DETAILED DESCRIPTION:
The study was conducted to describe and compare the plasma pharmacokinetics of NRL972 after a 15-second intravenous (i.v.) injection of 2 mg NRL972 against the diagnostic assessment based on liver biopsy in patients with clinically suspected NAFLD. A particular focus was to separate simple fatty liver disease (non-NASH) from non-alcoholic steatohepatitis (NASH) with or without cirrhosis (defined as advanced fibrosis: ≥F3) in a population likely to present with NAFLD.

The study evaluated the predictive value of NRL972 pharmacokinetics in the diagnosis of NASH using fatty liver disease (non-NASH) as the comparator group in a population of clinically suspected NAFLD patients based on histological evaluation. The sensitivity and specificity of NRL972 pharmacokinetics as a diagnostic was compared to that of results from the standard laboratory tests, clinical features, elastography assessments for liver stiffness and tests of metabolic markers, serum fibrosis markers and established disease scores frequently used in the evaluation of NAFLD.

The study also provided information on the safety and tolerability of i.v. doses of NRL972 under these conditions.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting the following conditions will be eligible for enrollment:

* Males or females (females of non-child-bearing potential or of child-bearing potential while taking medically appropriate contraception)
* Any ethnicity
* Age: 18 to 80 years of age
* Clinical evidence of non-alcoholic liver disease requiring the conduct of a liver biopsy for the diagnosis of NAFLD and/or staging of disease severity
* Willing and able to provide informed consent

Exclusion Criteria:

Subjects fulfilling any of the following criteria will be excluded from enrollment:

General - all subjects

* Presence of acute or chronic viral hepatitis confirmed by serology
* Clinical signs of significant cholestasis
* Liver impairment due to space-occupying processes (e.g. carcinoma)
* Liver transplant recipient or patient scheduled for liver transplantation
* Clinically evident rapidly deteriorating hepatic function
* Significant bleeding diathesis
* Esophageal bleeding within the 8 weeks prior to study entry
* Presence of any contraindications for the conduct of the planned liver biopsy (e.g. allergy to lidocaine, coagulopathy with <100 x109/L thrombocytes and/or INR >1.3
* History of any allergic reaction to fluorescein
* Presence of any acute infection
* Previous participation in this trial
* Having received any investigational drug or treatment within 30 days prior to study entry or requiring a concurrent treatment with any other experimental drug or treatment
* Uncontrolled hypo- or hypertension (treated or untreated) with resting systolic blood pressure >160 or < 90 mmHg, diastolic blood pressure >95 or < 50 mmHg
* Clinically relevant abnormal laboratory values indicating end-stage renal, pulmonary or cardiac disease
* Known HIV infection
* Concurrent alcohol use of more than 14 drinks (140g ethanol) for men and 7 drinks (70g ethanol) for women per week (each drink is counted as 10g ethanol)
* History of drug or alcohol abuse within 2 months prior to dosing
* Use of prohibited medication (section 4.8)
* Donation of blood during the last 60 days or a history of blood loss exceeding 300 mL within the last 3 months
* Suspicion or evidence that the subject is not trustworthy and reliable
* Suspicion or evidence that the subject is not able to make a free consent or to understand the information in this regard
* Significant side effects prior to the liver biopsy (e.g. anxiety requiring pre-medication) or after the biopsy (e.g. pain requiring i.v. pain medication, bleeding re-quiring medical intervention)

General - all females

* Positive pregnancy test
* Pre-menopausal women not using appropriate contraception

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2008-06; Primary Completion 2010-03 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
C(30)/C(10) | 30 minutes post-dose
  The primary efficacy variable was the NRL972 fractional retention ratio for 10 and 30 minutes post-dose (C30/C10) for different populations with NAFLD.
Adverse Events | Up to 2 hours post-dose
  Primary safety assessment: Incidence of treatment-emergent adverse events
Vital Signs | Up to 2 hours post-dose
  Primary safety assessment: continuous monitoring on automated cardiovascular systems

SECONDARY OUTCOMES:
C(60) | 60 minutes post-dose
  NRL972 fractional retention ratio for 60 minutes post-dose for different populations with NAFLD.
t1/2 | 60 minutes post-dose
  apparent terminal disposition half-life
CL | 60 minutes post-dose
  approximate overall clearance

CONTACTS AND LOCATIONS:
Overall Officials: Manal F Abdelmalek, M.D., MPH, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Glass O, Henao R, Patel K, Guy CD, Gruss HJ, Syn WK, Moylan CA, Streilein R, Hall R, Mae Diehl A, Abdelmalek MF. Serum Interleukin-8, Osteopontin, and Monocyte Chemoattractant Protein 1 Are Associated With Hepatic Fibrosis in Patients With Nonalcoholic Fatty Liver Disease. Hepatol Commun. 2018 Sep 21;2(11):1344-1355. doi: 10.1002/hep4.1237. eCollection 2018 Nov. PMID 30411081